CLINICAL TRIAL: NCT07196813
Title: Evaluation Of The Relationship Between Weaning Process And Delirium
Brief Title: The Association Between the Extubation Process and Delirium in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, ilker uğurlu, doctor, Eskisehir Osmangazi University
Other Study IDs: E-80558721-050.99-328825
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Delirium in the Intensive Care Unit; Mechanical Ventilation Complication
Keywords: delirium, CAM*ICU, PaO2/FiO2
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are limited studies in the literature investigating the relationship between delirium and the pre- and post-extubation periods in patients planned for extubation. Determining the impact of existing delirium during the extubation process or the possible causes of delirium occurring in this period may contribute to early recognition, prevention, or treatment of delirium. In our study, we screened patients scheduled for extubation in the intensive care unit using the Confusion Assessment Method for the ICU (CAM-ICU) before extubation and during the 48-hour post-extubation period to investigate the type of delirium, its relationship with sedation, and possible triggering and risk factors.

Methods: The study was conducted with 38 patients over 18 years old who had been on mechanical ventilation (MV) for at least 24 hours and had Richmond Agitation and Sedation Scale (RASS) scores between +4 and -3. CAM-ICU was applied to patients before extubation, and then the patients were weaned from mechanical ventilation. Age, sex, APACHE-II, SOFA, mCCI scores, length of stay, and duration of intubation were compared between CAM-ICU negative and positive patients before extubation, and the relationship with sedation type was evaluated. CAM-ICU was also applied at 24 and 48 hours after extubation, and the results were compared with arterial blood gas parameters including PaO2/FiO2, PCO2, and lactate levels.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were patients aged over 18 years, followed under MV for at least 24 hours, with a Richmond Agitation and Sedation Scale (RASS) score between +4 and -3, and for whom an extubation decision had been made

Exclusion Criteria:

* Exclusion criteria were patients with RASS scores of -4 or -5, patients with a history of neurocognitive disorders (dementia, Alzheimer's disease), and patients whose relatives did not provide consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study was carried out in patients who were followed under MV and in whom a decision for extubation was made by the attending physician. The sample size was determined as 38 patients
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The association between delirium and the 24-hour period before extubation and the 48-hour period after extubation in 38 patients for whom extubation was indicated. | Patient assessments were conducted during the period immediately before extubation and within the 48-hour period following extubation
  The study was carried out in patients who were followed under MV and in whom a decision for extubation was made by the attending physician. The sample size was determined as 38 patients. Delirium screening was performed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) during the period immediately before extubation and within the 48-hour period after extubation. In sedated patients, the sedative agent was recorded, and sedation was gradually reduced and discontinued 4-6 hours before each assessment. Immediately before extubation, the RASS was applied to assess the level of sedation and agitation. Patients with RASS scores between +4 and -3 were assessed using the CAM-ICU. At 24 and 48 hours after extubation, RASS was applied first, followed by CAM-ICU. Patients with a positive CAM-ICU result were considered to have delirium. The delirium subtype was determined according to the RASS score

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University Hospital, Eskişehir, Turkey (Türkiye)